CLINICAL TRIAL: NCT00239616
Title: Open-label Multicenter, Pharmacokinetic Study of a Single Dose of Intravenous Iron Sucrose in Adolescents on Hemodialysis or Peritoneal Dialysis Receiving Epoetin
Brief Title: Pharmacokinetic of Intravenous Iron Sucrose in Adolescents on Hemodialysis or Peritoneal Dialysis Receiving Epoetin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN01016
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; Pharmacokinetics
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron Sucrose (Experimental): A single 100 mg dose (1 vial), 20 mg/min injected over 5 minutes
  Interventions: Drug: Iron Sucrose injection

INTERVENTIONS:
Drug: Iron Sucrose injection — Iron sucrose 100 mg dose
  Other Names: Venofer

SUMMARY:
This is an open-label, multicenter pharmacokinetic study of Hemodialysis (HD) or Peritoneal Dialysis (PD) patients receiving erythropoietin. Patients were administered 100mg of iron sucrose undiluted by slow IV push over 5 minutes. Patients underwent serial blood draws and were subsequently followed for 7 days for safety endpoints.

DETAILED DESCRIPTION:
This is an open-label, multicenter pharmacokinetic study of HD of adolescent PD patients receiving erythropoietin. Patients between the ages of 12 and 18 were administered 100mg of iron sucrose, undiluted by slow IV push over 5 minutes, and underwent serial blood draws. The patients were subsequently followed for 7 days for safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 18 years
* History of Chronic Renal Failure requiring HD or PD
* Hgb </= 13 g/dL
* Ferritin < 800 ng/ml
* Transferrin Saturation (TSAT) < 50%
* Receiving epoetin

Exclusion Criteria:

* Known Sensitivity to Iron Sucrose
* Severe Concomitant disease of the liver or cardiovascular system
* Serious bacterial Infection
* Pregnancy / Lactation
* Active Hepatitis
* Patients with Causes of iron deficiency other that Chronic Renal Failure
* Blood Transfusion
* Body Weight < 25 kilograms
* Currently being treated for Asthma
* Received investigational drug within last 30 days

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2002-06-05 (Actual); Primary Completion 2003-09-15 (Actual); Study Completion 2003-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum Measured Plasma Concentration (Cmax) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Area Under the Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC 0-t) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; AUC 0-t is defined as AUC from time 0 to the last data point
Area Under the Curve From Time Zero Extrapolated to Infinity (AUC 0-∞) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC 0-∞ is defined as area under the concentration vs. time curve from zero to infinity.
Terminal Elimination Half-life (T1/2) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  T1/2 refers to the time taken for concentration of a drug to decrease from its maximum concentration to half of Cmax

SECONDARY OUTCOMES:
Total Body Clearance (CL) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  CL refers to the Dose/AUC 0-∞
Volume of Distribution (Vd) | 0, 5, 15, 30, 60, 90, 120, 240, 360, 480, and 720 minutes
  Vd refers to the ratio of amount of drug in a body (dose) to concentration of the drug that is measured in blood, plasma, and un-bound in interstitial fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.